CLINICAL TRIAL: NCT05503472
Title: Study Strategies in Musicians and Their Relationship With Respect to Musculoskeletal Status, Motivation and Artistic Level
Brief Title: Study Strategies in Musicians and Their Relationship With Physical and Emotional Variables
Acronym: SSMmusic
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Other Study IDs: ID0036
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Music
Keywords: Musicians; Musculoskeletal Pain; Strategies of study; Motivation and physiotherapy
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — observational

SUMMARY:
The musician profession requires great efforts not only at job level, also social, mental and physical level from the beginning of musical studies.

This study investigates the importance and the relationship between the strategies of study, the artistic level and the motivational level in prevalent musculoskeletal diorders in music students.

The aim of this study is to check the different areas that can influence study strategies, the importance of motivation, music students' deficiencies and assess the contribution of physiotherapy during music studies. To do this, a questionnaire will be sent to students from different conservatories and master's degrees.

DETAILED DESCRIPTION:
Most of the musicians' careers start from childhood, and the demands on both the physical and psychosocial levels entail a large number of occupational diseases and risks to their health. Music students need to dedicate a significant number of hours per day in their different stages of their musical career if they want to achieve success in the studio and turn their studies into their future profession. To meet their objectives, aspects such as motivation, support and adopting good study strategies, among others, are necessary.

The psychological as well as social and physical factors that influence the professional life of the musician. Therefore, working on them from the beginning of the studies, with good practices and strategies, can lead them to success. However, having real information on music students and knowing these aspects would allow us to know the real extent of the motivation and study strategies that the student proposes to improve their musical practice, the discomfort or muscle pain they suffer and the relationship between all of them. Therefore, it is necessary to know the study strategies applied by music students, as well as to know the motivation and how it can affect musical practice and relate to muscular discomfort so frequent in this population group. The main objective of this study is to know the study strategies of conservatory music students, their artistic and motivational level and the possible relationship with musculoskeletal disorders.

Study design. The type of study is a cross-sectional descriptive study that will be carried out through an online questionnaire using the Google Forms platform specially designed for this study. The participating subjects voluntarily, guaranteeing the confidentiality and anonymity of the study participants, as well as their responses. By accessing the questionnaire, the subject has been informed about the purpose and purpose of the study and has given their consent.

This study investigates the importance and the relationship between the strategies of study, the artistic level and the motivational level in prevalent musculoskeletal diorders in music students.

ELIGIBILITY:
Inclusion Criteria:

* Be a music student, either master's or conservatory
* Being over 18 years
* Study an instrument or song

Exclusion Criteria:

* Not studying or having studied any music course
* Be under 18 years of age

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Music student
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Study quality | 1 day
  This section is elaborated with specific questions for the present study, it asks about the study time per day in hours, the complete days of weekly rest, you spend in the daily study (duration of the breaks and criteria to make a break), use of the metronome, recordings to listen to and make corrections, visualization exercises, time planning, form and content of study, setting objectives per session: obtaining better results.

SECONDARY OUTCOMES:
Self-care and Musculoskeletal Status | 1 day
  Regarding self-care and musculoskeletal status, they elaborate specific questions for the present study. Data are obtained regarding previous warm-up exercises and final stretching exercises, mode of action against muscular discomfort, the type of muscular pain and the specific area of pain (back, upper limb or lower limb), fear when playing sports, daily continuous exercise for more than 30 min, days of exercise/week and type of exercise performed and the subject's physical state.
Mood | 1 day
  It consists of specific questions for the present study, including questions about the feelings that students present when playing an instrument, the joy or motivation that it causes them or the level of frustration that they can reach when making a mistake.
Motivational level | 1 day
  Motivational level It consists of work with specific questions for this study, information is collected about the family support they receive during their studies in music, the level as a performer they consider to have and the score received in the last course.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma Espí, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No